CLINICAL TRIAL: NCT01613586
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Parallel Group, Adaptive, Combined Proof of Concept and Dose-Finding Study to Investigate Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of ASP3652 in the Treatment of Female Patients With Bladder Pain Syndrome / Interstitial Cystitis
Brief Title: A Randomized Study Comparing Placebo and ASP3652 in the Treatment of Women With Bladder Pain Syndrome / Interstitial Cystitis (BPS/IC)
Acronym: AMARANTH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3652-CL-0018; 2011-004555-39 (EudraCT Number)
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Cystitis, Interstitial; Urinary Bladder Disease; Pain; Urologic Diseases
Keywords: ASP3652; Painful Bladder Syndrome; Interstitial Cystitis; Bladder Pain Syndrome
MeSH Terms: conditions — Cystitis, Interstitial; Urinary Bladder Diseases; Pain; Urologic Diseases | interventions — ASP3652

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose ASP3652 twice daily (Experimental): 50 mg twice daily for 12 weeks
  Interventions: Drug: ASP3652
- Medium dose ASP3652 twice daily (Experimental): 150 mg twice daily for 12 weeks
  Interventions: Drug: ASP3652
- High dose ASP3652 twice daily (Experimental): 300 mg twice daily for 12 weeks
  Interventions: Drug: ASP3652
- Placebo (Placebo Comparator): Matching placebo twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP3652 — Oral
  Arms: High dose ASP3652 twice daily; Low dose ASP3652 twice daily; Medium dose ASP3652 twice daily
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
In this study several dose levels of ASP3652, given orally for 12 weeks, will be compared with placebo in the treatment of female patients with Bladder Pain Syndrome / Interstitial Cystitis.

DETAILED DESCRIPTION:
This study consists of a screening phase, an initial 3 weeks Run-in period,

a 12 weeks Treatment period and a 2 weeks Follow-up (FU) period.

This study will investigate the efficacy and safety of a 12 week treatment with ASP3652 in female patients with Bladder Pain Syndrome / Interstitial Cystitis (BPS/IC). Different dose levels of ASP3652 will be compared with placebo. ASP3652 is administered as oral tablets. The objectives of the study are to investigate efficacy of ASP3652 in patients with BPS/IC, to assess the optimal dose of ASP3652, to investigate safety and tolerability and to investigate pharmacokinetics and pharmacodynamics of ASP3652 in patients with BPS/IC in an out-patient setting.

ELIGIBILITY:
Inclusion Criteria:

* Has previously been diagnosed with BPS/IC; i.e., pelvic pain, pressure or discomfort perceived to be related to the urinary bladder accompanied by at least one other urinary symptom such as persistent urge to void or frequency, for at least 3 months prior to screening in absence of urinary infection or other obvious pathology or identifiable causes
* Has at enrolment a score of 4 or greater on the 11-point (0-10) NRS for average pain over the previous week, which is item 4 of the F-GUPI
* Has a mean pain score of 4.0 or greater on the 11-point (0-10) NRS for daily assessed pain (item 4 of F-GUPI-24H) over the last 7 days prior to randomization
* Is willing to comply with study requirements such as completing the questionnaires and diaries and attend all study visits and practicing birth control

Exclusion Criteria:

* Undergone a cystoscopy with hydrodistension or undergone Botox injections in the bladder within 6 months prior to screening
* Use of pentosan polysulphate sodium within 4 weeks prior to screening
* Any intravesicular pharmacological treatment or other interventions for BPS/IC or bladder, urethral, ureteral, pelvic or peri-pelvic invasive procedure within 3 months prior to screening
* Cystitis or documented symptomatic bacterial cystitis in the last 3 months prior to screening
* Lower urinary tract malignancy, such as positive (micro) hematuria in urine sediment
* Neurologic disease or defect affecting bladder function or symptomatic urethral diverticulum or any post-partum or surgery related genital tract conditions, symptomatic bladder or ureteral calculi or Post Void Residual volume greater than 150 mL
* Clinically significant abnormalities observed during cystoscopy or on transabdominal ultrasound
* Currently active or treated sexual transmittable diseases
* Substance abuse or any use of delta-9-tertrahydrocannabinol (THC) as assessed by a positive urine test for THC at screening
* Any clinically relevant concomitant disease (past or present) which would, in the opinion of the investigator, put the subject at risk or mask measures of efficacy
* Symptoms of depression, defined as a Center for Epidemiological Studies Depression Scale score of 27 or more
* Use of steroids, immunomodulators, cytochrome P4502C8 inhibitors, cannabis / THC based medication, opioid analgesics or antiviral / antibacterial / antifungal agents during the last 4 weeks before the screening
* Initiation, discontinuation, or variation in the dose of antidepressants, anticonvulsants, antimuscarinics, benzodiazepines, skeletal muscle relaxants, non-steroid anti-inflammatory drugs, non opioid analgesics, homeopathic medication and herbal therapies during the last 4 weeks before the screening. Subjects should continue these medications at that same stable dose throughout the study
* Clinically relevant abnormal urine or blood safety laboratory values or active hepatic and/or biliary disease (AST or ALT should not be >2 times the upper limit of normal, total bilirubin should not be >1.5 times the upper limit of normal)
* Participated in any clinical study or has been treated with any investigational drug or device within 84 days or the period stipulated by local regulations, whichever is longer, prior to the screening

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2012-05-31 (Actual); Primary Completion 2014-03-18 (Actual); Study Completion 2014-03-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Mean Daily Pain (MDP) at 12 weeks | Baseline and 12 weeks
  Pain is assessed on an 11 point (0-10) Numerical Rating Scale (NRS), which is item 4 of the Female GenitoUrinary Pain Index (24 hours recall) (F-GUPI-24h)

SECONDARY OUTCOMES:
Change from baseline in Mean Daily Pain (MDP) at 4, 8 weeks treatment and at 2 weeks follow-up post treatment | Baseline, 4 and 8 weeks treatment and 2 weeks follow-up post treatment
  Pain is assessed on an 11 point (0-10) Numerical Rating Scale (NRS), which is item 4 of the F-GUPI-24h
Change from baseline in Female GenitoUrinary Pain Index (one week recall) (F-GUPI) Total score at 4, 8, 12 weeks treatment and at 2 weeks follow-up post treatment | Baseline, 4, 8, 12 weeks treatment and 2 weeks follow-up post treatment
Change from baseline in F-GUPI Pain subscale score, Urinary subscale score, and Quality of Life Impact score at 4, 8, 12 weeks treatment and at 2 weeks follow-up post treatment | Baseline, 4, 8, 12 weeks treatment and at 2 weeks follow-up post treatment
Daily pain, assessed with item 4 of the F-GUPI-24h during Run-in, Treatment period and Follow-up post treatment | Every day during the Run-in, Treatment and Follow-up post treatment periods
Change from baseline in questionnaires at 12 weeks treatment | Baseline and 12 weeks treatment
  Bladder Pain/IC Symptom Score; O'Leary-Sant IC Symptom & Problem Index; Short form McGill pain questionnaire; Female Sexual Function Index; European Quality of Life questionnaire in 5 Dimensions
Global Response Assessment (GRA) at 0, 4, 8 and 12 weeks treatment and at 2 weeks follow-up post treatment | Baseline, 4, 8, 12 weeks treatment and 2 weeks follow-up post treatment
  GRA is assessed as change from baseline which is here start of Run-in period
Change from baseline in Voiding parameters (urinary frequency, urinary urgency, nocturia and total urgency score ) at 4, 8, 12 weeks treatment and at 2 weeks Follow-up post treatment | Baseline, 4, 8, 12 weeks treatment and 2 weeks follow-up post treatment
Proportion of responders: at least 7-point decrease in F-GUPI Total score at 0, 4, 8 and 12 weeks treatment compared to baseline | Baseline, 4, 8 and 12 weeks treatment
Assessment of pharmacokinetics at week 4, 8 and 12 | 4, 8 and 12 weeks treatment
  Plasma levels of ASP3652
Assessment of pharmacodynamics at week 4, 8 and 12 | 4, 8 and 12 weeks treatment
  Plasma levels of anandamides
Safety as assessed by recording Adverse Events, Laboratory tests, electrocardiograms (ECGs) and vital signs | Baseline and 12 weeks treatment
Safety as assessed by SteatoTest, adiponectin and PVR | Baseline and 12 weeks
Change from baseline in questionnaires (Center for Epidemiologic Studies Depression Scale and Profile of Mood States questionnaire) at 12 weeks treatment | Baseline and 12 weeks treatment
Physician Withdrawal Checklist at 12 weeks treatment and at 2 weeks follow-up post treatment | 12 weeks treatment and 2 weeks follow-up post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Director — Astellas Pharma Europe B.V.
Locations (60):
- Belgium (2):
  - Site: 5101, Antwerp
  - Site: 5103, Brussels
- Czechia (6):
  - Site: 5202, Kralove
  - Site: 5203, Kroměříž
  - Site: 5206, Olomouc
  - Site: 5209, Pilsen
  - Site: 5210, Sternberk
  - Site: 5201, Uherské Hradiště
- Denmark (3):
  - Site: 5303, Aarhus
  - Site: 5301, Herlev
  - Site: 5302, Næstved
- Germany (8):
  - Site: 5406, Duisburg
  - Site: 5403, Emmendingen
  - Site: 5409, Frankfurt am Main
  - Site: 5402, Holzminden
  - Site 5410, Kirchheim
  - Site: 5405, Mainz
  - Site: 5404, Nürtingen
  - Site: 5414, Offenburg
- Latvia (3):
  - Site: 5602, Liepāja
  - Site: 5601, Riga
  - Site: 5603, Riga
- Lithuania (4):
  - Site: 6304, Kaunas
  - Site: 6302, Vilnius
  - Site: 6301, Vilnius
  - Site: 6303, Vilnius
- Netherlands (5):
  - Site: 5706, Amsterdam
  - Site: 5703, Maastricht
  - Site: 5701, Nijmegen
  - Site: 5702, Winterswijk
  - Site: 5704, Zwijndrecht
- Poland (9):
  - Site: 5807, Bialystok
  - Site 5806, Bydgoszcz
  - Site: 5811, Chorzów
  - Site: 5801, Lodz
  - Site: 5805, Piaseczno
  - Site: 5812, Poznan
  - Site: 5802, Warsaw
  - Site: 5804, Warsaw
  - Site: 5803, Warsaw
- Portugal (3):
  - Site 5902, Coimbra
  - Site 5903, Porto
  - Site 5901, Porto
- Romania (7):
  - Site 6006, Brasov
  - Site 6003, Bucharest
  - Site 6004, Bucharest
  - Site 6007, Bucharest
  - Site 6002, Bucharest
  - Site 6005, Iași
  - Site 6001, Târgu Mureş
- Russia (6):
  - Site 6108, Moscow
  - Site 6103, Moscow
  - Site: 6111, Moscow
  - Site 6106, Moscow
  - Site 6101, Moscow
  - Site 6102, Saint Petersburg
- Spain (4):
  - Site 6202, Laguna, Tenerife
  - Site 6203, Barcelona
  - Site 6201, Barcelona
  - Site 6204, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=287